CLINICAL TRIAL: NCT07199673
Title: Comparison of Outcome of Injection Sclerotherapy Versus Rubber Band Ligation for Second Degree Hemorrhoids
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulab Devi Hospital (Other)
Responsible Party: Principal Investigator, Mudassar Malik, Post Graduation Resident, Gulab Devi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAMC/IRB/EA252025
Record Dates: First submitted 2025-09-19; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hemorrhoid
Keywords: Injection Sclerotherapy; Rubber Band Ligation; Second Degree Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group IST (Other): 5% phenol in almond oil
  Interventions: Drug: Injection Sclerotherapy
- Group RBL (Other): rubber band is applied at the base of each hemorrhoid using Barron's Gun and Elise's tissue forceps.
  Interventions: Device: Rubber Band Ligation

INTERVENTIONS:
Drug: Injection Sclerotherapy — identifying the hemorrhoidal pedicle, 3-5 ml of 5% phenol in almond oil is injected into the submucosal plane of the hemorrhoid pedicle
  Arms: Group IST
Device: Rubber Band Ligation — knee-elbow position is used. After identifying the hemorrhoids with a proctoscope, a rubber band is applied at the base of each hemorrhoid using Barron's Gun and Elise's tissue forceps.
  Arms: Group RBL

SUMMARY:
Objective of this study is to compare the outcome of Injection Sclerotherapy versus Rubber Band Ligation for second degree hemorrhoids in terms of bleeding and efficacy.

DETAILED DESCRIPTION:
There is a difference in the outcome of Injection Sclerotherapy versus Rubber Band Ligation for second degree hemorrhoids in terms of bleeding and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 75 who have been diagnosed with second-degree hemorrhoids

Exclusion Criteria:

* Patients with thrombosed hemorrhoids, and those with serious comorbid conditions such as heart, kidney, or liver diseases, coagulation disorders, or severe anemia.

  * Individuals who have received treatment for hemorrhoids in the past six months.
  * Pregnant women.
  * Patients unable to commit to necessary follow-up appointments.
  * Patients with a history or current presence of colorectal cancer or anal malignancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-01-06 (Estimated); Study Completion 2026-01-06 (Estimated)

PRIMARY OUTCOMES:
Early per rectal Bleeding | 24 hours
  within 24 hours post-procedure

SECONDARY OUTCOMES:
Delayed Bleeding Per rectal | 24 hours to 14th post operative day
  24 hours to 14th post-operative day

CONTACTS AND LOCATIONS:
Locations (1):
- Gulab devi Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
i am collecting my data for study. I did not completed my data. so i am unable to share